CLINICAL TRIAL: NCT02220621
Title: A Prospective, Multi-center, Randomized, Controlled Clinical Study on Self-crosslinked Sodium Hyaluronate Gel for Prevention of Intrauterine Adhesion
Brief Title: Efficacy and Safety of Crosslinked Hyaluronan Gel for Preventing Intrauterine Adhesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaozheng Shu (Industry)
Responsible Party: Sponsor-Investigator, Xiaozheng Shu, CEO, BioRegen Biomedical (CHangzhou) Co., Ltd
Organization: BioRegen Biomedical (CHangzhou) Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FNL-2011-03
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Intrauterine Adhesion
Keywords: Intrauterine adhesion; crosslinked hyaluronan gel; hysteroscopy; clinical trial
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Treatment (Experimental): After the hysteroscopic adhesiolysis, crosslinked hyaluronic acid gel is applied into the uterine cavity, then a Foleys balloon catheter is inserted into the uterine cavity.
  Interventions: Device: Crosslinked hyaluronic acid gel; Device: Foleys balloon catheter
- Control (Active Comparator): After hysteroscopic adhesiolysis, a Foleys balloon catheter is inserted into the unterine cavity.
  Interventions: Device: Foleys balloon catheter

INTERVENTIONS:
Device: Crosslinked hyaluronic acid gel — After hysteroscopic adhesiolysis, MateRegen Gel IU is applied into the uterine cavity together with a Foley balloon catheter.
  Other Names: MateRegen Gel IU.
  Arms: Treatment
Device: Foleys balloon catheter — After adhesivolysis, the Foleys balloon catheter is inserted into the uterine cavityand expanded with normal saline.

SUMMARY:
Intrauterine adhesion (IUA) is the adhesion of intrauterine tissues due to the exposure of myometrial tissues caused by the endometrial basal injury. IUA is clinically manifested as symptoms such as abdominal pain, hypomenorrhea or amenorrhea, sterility and habitual abortion, which seriously affect the patients quality of life.

Preventing IUA has been tried using different methods such as barrier or stent in order to separate the opposing endometrium during the tissue healing processes. Although some successes have been reported there are still some challenges need to be dealt with.

One of the barrier materials for preventing IUA is made of hyaluronic acid (HA). HA is a natural ECM of human tissue with excellent biocompatibility and promotes the scar-free wound repair. The self-crosslinked esterified HA gel has demonstrated the capacity to prevent IUA in clinical studies.

A novel self-crosslinked HA gel is developed by BioRegen Biomedical（Changzhou）Co., Ltd with proprietary technologies. This product is a highly viscoelastic crosslinked gel that overcomes the shortcoming of sodium hyaluronate with high motility and too quick degradation in vivo. For this product, the results of animal experiments and various safety features have been designed and tested conforming to the national regulations and standards. In order to launch this product to the market, this prospective, randomized and controlled clinical trial is designed and will be performed to verify its safety/efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients who are 20-40 years old who is diagnosed as intrauterine adhesion, and did not receive adhesiolysis surgery.
* Patients who signed the informed consent form (ICF) and agreed to take contraceptive measures within 3 months after the surgery.
* Physical examination and routine laboratory tests demonstrated no systemic diseases.
* According to the AFS scoring system on the IUA (1988) only those patients with moderate to severe IUA (i.e. total AFS score larger than 4 points) were enrolled in this clinical trial.

Exclusion Criteria:

* Patients who is allergic to hyaluronan or its derivatives.
* Patients with inflammation of reproductive organs, pelvic cavity inflammation, malignant tumor of reproductive organs and other systemic diseases that could cause metrorrhagia.
* Patients with malformation of reproductive organs.
* Patients who may not take effective contraceptive measures within 3 months after the surgery. Patients who were suffering severe systemic diseases such as coagulative disorders, cardiovascular diseases and long-term alcoholism and drug abuse were also excluded from this clinical trial.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
the percentage of patients free from IUA | 3 months after surgery
  Second look hysteroscopic examinations were performed at 3 months postoperatively. The adhesion was scored at adhesiolysis surgery and at follow-up hysteroscopy according to American Fertility Society scoring system.

SECONDARY OUTCOMES:
Effective rate | three months after surgery
Total AFS score | 3 months
The score for each subcategory of AFS scoring system | 3 months
The safety | 3 months
  Evaluated based on the number of patients shown complications and incidence rate for severe adverse events

OTHER OUTCOMES:
Safety | 3 months
  Severe adverse event (SAE): cause prolonged hospitalization and disability to the patient.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The People's Hospital of Hunan Province, Changshu, Hunan
  - The People's Hospital of Chenzhou City,, Chenzhou, Hunan

REFERENCES:
- [Background] Acunzo G, Guida M, Pellicano M, Tommaselli GA, Di Spiezio Sardo A, Bifulco G, Cirillo D, Taylor A, Nappi C. Effectiveness of auto-cross-linked hyaluronic acid gel in the prevention of intrauterine adhesions after hysteroscopic adhesiolysis: a prospective, randomized, controlled study. Hum Reprod. 2003 Sep;18(9):1918-21. doi: 10.1093/humrep/deg368. PMID 12923149